CLINICAL TRIAL: NCT00884065
Title: Effectiveness of Diacutaneous Fibrolysis on Pain and Mobility in Patients Suffering From Painful Shoulder. A Randomized Pilot Study.
Brief Title: Effectiveness of Diacutaneous Fibrolysis in Painful Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Idiap08/187
Record Dates: First submitted 2009-02-09; First posted 2009-04-20 (Estimated); Results first posted 2009-04-20 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Shoulder Pain
Keywords: Physiotherapy; Manual therapy; Painful Shoulder; Diacutaneous Fibrolysis
MeSH Terms: conditions — Shoulder Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Intervention Group (Experimental): The intervention group was treated with a single session of DF following the procedure as described by the authors.
  Interventions: Other: Diacutaneous Fibrolysis
- Control Group (Placebo Comparator): The control group was treated with a single placebo session of DF.
  Interventions: Other: Diacutaneous Fibrolysis (placebo)

INTERVENTIONS:
Other: Diacutaneous Fibrolysis — The implementation of the technique consists of three consecutive stages: The first stage involves manual palpation, which is carried out by the hand that is not holding the hook, with the objective to find the area to be treated; the second, or instrumental palpation stage, is carried out by introducing the spatula of the hook together with the index finger of the palpatory hand to locate with precision the adherent connective fibers or fibrous corpuscles; the third, or fibrolysis stage, is the actual treatment. Here, a brief supplementary traction is carried out with the hook.
  Other Names: Manual therapy
  Arms: Intervention Group
Other: Diacutaneous Fibrolysis (placebo) — The placebo was designed for this study and the stages of manual and instrumental palpation occur strictly at a superficial level. In the third stage, instead of fibrolysis a pinch of skin is hold with the thumb of the palpatory hand and the tip of the spatula, so that the patient feels the hook distinctly but without any action taking place on the deep tissular planes.
  Other Names: Manual therapy
  Arms: Control Group

SUMMARY:
While Diacutaneous fibrolysis (DF) has achieved promising results empirically, its effectiveness has not been tested in clinical trials. The investigators hypothesized that the use of DF in patients suffering from painful shoulder would increase the active mobility and reduce the pain during movement. To test the hypothesis a double blind (patient and investigator) randomized clinical trial was carried out in two public Primary Health Care Centres. Fifty patients were randomly allocated to two groups: the intervention group, who received a real DF session, and the control group, who received a placebo DF session.

DETAILED DESCRIPTION:
Background and objectives:

Diacutaneous fibrolysis (DF) is a manual technique to treat the mechanical pain of the musculoskeletal system. While this technique has achieved promising results empirically, its effectiveness has not been tested in clinical trials. We aimed at evaluating the effectiveness of a single session of DF on pain and mobility in patients suffering from painful shoulder.

Subjects and methods:

This clinical trial took place in two public Primary Health Care Centres. Fifty patients were randomly allocated to two groups: the intervention group, who received a real DF session, and the control group, who received a placebo DF session. The degree of active mobility (flexion, abduction, extension, external and internal rotation), the pain in the hand behind back position and the participant's perception of the technique in terms of comfort and results obtained were measured.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* being referred for treatment of painful shoulder (except for adhesive capsulitis)
* not having been previously treated with DF

Exclusion Criteria:

* Damaged skin and/or cutaneous lesions in the shoulder area
* History of shoulder surgery
* Vascular abnormalities
* Platelet antiaggregant therapy
* Acute inflammatory condition of the shoulder (<1 week)
* Patients with a pending litigation or court claim

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martín-Eusebio Barra-López, PT, Principal Investigator — Catalan Institute of Health; Carlos López-de-Celis, DO, PT, Principal Investigator — Catalan Institute of Health; Gabriela Fernández-Jentsch, PT, Principal Investigator — Servicio Gallego de Salud; Ernesto Murillo-Barrios, PT, Principal Investigator — Servicio Gallego de Salud; Edurne Villar-Mateo, PT, Principal Investigator — Catalan Institute of Health; Laura Raya-de-Cardenas, PT, Principal Investigator — Catalan Institute of Health
Locations (1):
- Catalan Institute of Health - Servei de Rhb Sant Ildefons, Cornellà de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Barra ME, Lopez C, Fernandez G, Murillo E, Villar E, Raya L. The immediate effects of diacutaneous fibrolysis on pain and mobility in patients suffering from painful shoulder: a randomized placebo-controlled pilot study. Clin Rehabil. 2011 Apr;25(4):339-48. doi: 10.1177/0269215510385480. Epub 2010 Nov 15. PMID 21078700

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were recruited from two public services of primary health care of the Spanish National Health Service, one in Cornellà de Llobregat (Barcelona), the other in Ponteareas (Pontevedra), from June 2007 to January 2008.
Groups:
- Intervention Group (Diacutaneous Fibrolysis): The intervention group was treated with a single session of Diacutaneous Fibrolysis following the standard procedure.
- Control Group (Placebo): The control group was treated with a single placebo session of Diacutaneous Fibrolysis.
Period: Overall Study
Arm/Group | Intervention Group (Diacutaneous Fibrolysis) | Control Group (Placebo)
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group (Diacutaneous Fibrolysis) | Control Group (Placebo) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 17 | 15 | 32.0
  >=65 years | 8 | 10 | 18.0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.76 (10.33) | 60.8 (10.12) | 58.78 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29.0
  Male | 9 | 12 | 21.0
Region of Enrollment [Number; unit: participants]
  Spain | 25 | 25 | 50.0
Months of pain [Mean (Standard Deviation); unit: Months] | 14.48 (16.21) | 17.88 (27.56) | 16.18 (22.44)

OUTCOME MEASURES:

1. Secondary Outcome: Change in Pain in the Hand Behind Back Position After Intervention Minus Baseline
Description: An unmarked Visual Analogue Scale from 0 (no pain) to 100 (worst pain) millimeters was used. At baseline, participants registered the pain perceived in the position used to measure the internal rotation. After intervention, they registered the pain with the hand placed in the same position taking as a reference the mark in the first evaluation.
Time Frame: Baseline and the same day (just after intervention)
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Intervention Group (Diacutaneous Fibrolysis) | Control Group (Placebo)
Number analyzed (Participants) | 25 | 25
Millimeters | -9.20 (15.16) | -7.48 (13.68)
Statistical Analysis 1: Comparison: Intervention Group (Diacutaneous Fibrolysis) vs Control Group (Placebo); Test type: Superiority or Other; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = -1.72, 95% CI 2-sided [-9.93 to 6.49], Standard Error of Mean 4.08

2. Primary Outcome: Change in Active Flexion Movement After Intervention Minus Baseline
Description: A universal double armed goniometer was used to measure change in active flexión movement in the sagital plane with the elbow fully extended and the forearm in indifferent pronosupination (thumb forward)
Time Frame: Baseline and the same day (just after intervention)
Measure: Mean (Standard Deviation); unit: Sexagesimal Degrees
Arm/Group | Intervention Group (Diacutaneous Fibrolysis) | Control Group (Placebo)
Number analyzed (Participants) | 25 | 25
Sexagesimal Degrees | 9.48 (10.86) | -1.92 (9.03)
Statistical Analysis 1: Comparison: Intervention Group (Diacutaneous Fibrolysis) vs Control Group (Placebo); Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 11.40, 95% CI [5.72 to 17.08], Standard Error of Mean 2.83

3. Primary Outcome: Change in Active Abduction Movement After Intervention Minus Baseline
Description: A universal double armed goniometer was used to measure change in active abduction movement in the scapular plane with the elbow in extension and the forearm in supination
Time Frame: Baseline and the same day (just after intervention)
Measure: Mean (Standard Deviation); unit: Sexagesimal degrees
Arm/Group | Intervention Group (Diacutaneous Fibrolysis) | Control Group (Placebo)
Number analyzed (Participants) | 25 | 25
Sexagesimal degrees | 7.88 (9.61) | 0.64 (8.69)
Statistical Analysis 1: Comparison: Intervention Group (Diacutaneous Fibrolysis) vs Control Group (Placebo); Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 7.24, 95% CI 2-sided [2.03 to 12.45], Standard Error of Mean 2.59

4. Primary Outcome: Change in Active extensión Movement After Intervention Minus Baseline
Description: A universal double armed goniometer was used to measure change in active extensión movement in the sagital plane with the elbow fully extended and the forearm in indifferent pronosupination (thumb forward)
Time Frame: Baseline and the same day (just after intervention)
Measure: Mean (Standard Deviation); unit: Sexagesimal degrees
Arm/Group | Intervention Group (Diacutaneous Fibrolysis) | Control Group (Placebo)
Number analyzed (Participants) | 25 | 25
Sexagesimal degrees | 2.08 (5.66) | 0.16 (6.44)
Statistical Analysis 1: Comparison: Intervention Group (Diacutaneous Fibrolysis) vs Control Group (Placebo); Test type: Superiority or Other; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 1.92, 95% CI 2-sided [-1.53 to 5.37], Standard Error of Mean 1.72

5. Primary Outcome: Change in Active External Rotation After Intervention Minus Baseline
Description: A universal double armed goniometer was used to measure change in active external rotation measured in the neutral position of the shoulder (arm pinned to the trunk), elbow flexed to 90º and the forearm in indifferent pronosupination (thumb forward)
Time Frame: Baseline and the same day (just after intervention)
Measure: Mean (Standard Deviation); unit: Sexagesimal degrees
Arm/Group | Intervention Group (Diacutaneous Fibrolysis) | Control Group (Placebo)
Number analyzed (Participants) | 25 | 25
Sexagesimal degrees | 0.76 (9.55) | 0.16 (5.24)
Statistical Analysis 1: Comparison: Intervention Group (Diacutaneous Fibrolysis) vs Control Group (Placebo); Test type: Superiority or Other; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [-3.81 to 5.01], Standard Error of Mean 2.18

6. Primary Outcome: Change in Active Internal Rotation After Intervention Minus Baseline
Description: Change in active internal rotation was measured with the hand behind back test. The position achieved by the tip of the thumb was marked and with a flexible metric tape (always the same) the distance in centimetres between this mark and the inferior tip of the spinous process of C7 was measured; the shorter the distance, the better the mobility
Time Frame: Baseline and the same day (just after intervention)
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Intervention Group (Diacutaneous Fibrolysis) | Control Group (Placebo)
Number analyzed (Participants) | 25 | 25
Centimeters | 4.50 (6.79) | 1.42 (3.12)
Statistical Analysis 1: Comparison: Intervention Group (Diacutaneous Fibrolysis) vs Control Group (Placebo); Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 3.08, 95% CI 2-sided [0.08 to 6.09], Standard Error of Mean 1.49

ADVERSE EVENTS:
Arm/Group | Intervention Group (Diacutaneous Fibrolysis) | Control Group (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No